CLINICAL TRIAL: NCT06122662
Title: A Phase 2b/3 Study of the Safety and Efficacy of AMX0035 in Progressive Supranuclear Palsy (ORION)
Brief Title: AMX0035 and Progressive Supranuclear Palsy
Acronym: ORION
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A35-009
Record Dates: First submitted 2023-11-03; First posted 2023-11-08 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Progressive Supranuclear Palsy; PSP; Neurodegenerative Diseases; Atypical Parkinsonism
Keywords: Progressive Supranuclear Palsy; PSP; Steele-Richardson-Olszewski Syndrome; ORION; Amylyx
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Neurodegenerative Diseases | interventions — sodium phenylbutyrate and taurursodiol

STUDY DESIGN:
Intervention Model Description: A35-009 (ORION) is a blinded, randomized, placebo-controlled, two-part Phase 2b/3 study, each part consisting of a 52-week double-blind, placebo-controlled phase followed by an optional 52-week open-label extension phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, Care providers, Investigators, and study staff will be blinded to participant group assignment during the double-blind phase and extension phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMX0035 (Experimental): AMX0035 administered by mouth for 52 weeks: once daily for first 2 weeks and then twice daily for remainder of study
  For participants electing to continue into the open-label phase at Week 52; AMX0035 will be administered once daily for first 2 weeks and then twice daily for remainder of open-label phase
  Interventions: Drug: AMX0035
- Placebo (Placebo Comparator): Placebo administered by mouth for 52 weeks: once daily for first 2 weeks and then twice daily for remainder of study
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AMX0035 — Proprietary formulation of sodium phenylbutyrate and taurursodiol
  Arms: AMX0035
Other: Placebo — Matching Placebo Comparator
  Arms: Placebo

SUMMARY:
A35-009 (ORION) is a Phase 2b/3 trial to evaluate the efficacy and safety of AMX0035 in participants with Progressive Supranuclear Palsy (PSP), consisting of randomized, double blind placebo controlled phases, followed by an optional open-label extension phase.

DETAILED DESCRIPTION:
AMX0035 is a fixed dose combination therapy designed to reduce neuronal death through blockade of key cellular death pathways originating in the endoplasmic reticulum (ER) and mitochondria. This clinical trial is designed to demonstrate that AMX0035 is safe and tolerable, and to assess its effect on disease progression as measured by the Progressive Supranuclear Palsy (PSP) Rating Scale (PSPRS) over a 52-week double-blind phase. The Phase 2b and Phase 3 study portions are planned to feature an identical design: a randomized, double-blind, placebo-controlled phase that is followed by an optional open-label extension (OLE) phase. The phase 3 portion of ORION may be initiated based on results of the phase 2b Interim Analysis and/or the Primary Analysis and the totality of data from the Phase 2b study portion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 40 to 80 years of age, inclusive
* Diagnosis of possible or probable PSP Richardson Syndrome
* Presence of PSP symptoms for <5 years
* Score of <40 on the total (28-item) Progressive Supranuclear Palsy Rating Scale (PSPRS)
* Able to walk independently or with minimal assistance
* Minimum score of 24 on the Mini Mental State Examination (MMSE)
* Must reside outside a skilled nursing facility or dementia care facility at the time of screening. Residence in an assisted living facility is allowed
* Must have a study partner willing to attend study visits and provide information on participant's status
* Capable of providing informed consent
* Capable and willing to comply with trial procedures including visits to the trial clinic, visit requirements and treatment schedule, including MRI scans
* Female participants of childbearing potential must agree to use effective birth control for the duration of the study and for 6 months after last dose of study drug.
* Males must agree to use effective birth control method for the duration of the study and for 6 months after the last dose of study drug. Men must not plan to donate sperm.

Exclusion Criteria:

* Require use of a feeding tube
* Evidence of any neurological disorder that could explain signs of PSP
* Evidence of any clinically significant neurological disorder other than PSP, including significant cerebrovascular abnormalities, vascular dementia, motor neuron disease or ALS, Huntington's disease, normal pressure hydrocephalus, brain tumor, seizure disorder, multiple sclerosis, or known structural brain abnormalities.
* History of autosomal dominant PSP due to a Microtubule Associated Protein Tau (MAPT) mutation
* History of an autosomal dominant mutation associated with Frontotemporal Lobar Degeneration (FTLD)
* Prior or current diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
* Presence of unstable psychiatric disease, cognitive impairment (e.g., major cognitive dysfunction), dementia, major depression, or substance abuse that would impair ability of the participant to provide informed consent and follow instructions
* Abnormal liver function
* Renal insufficiency
* Ongoing anemia
* History of Class III/IV heart failure per New York Heart Association (NYHA)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in total (28-item) Progressive Supranuclear Palsy Rating Scale (PSPRS) Score | 52 weeks
  Assess the impact of AMX0035 on disease progression as measured by the Progressive Supranuclear Palsy (PSP) Rating Scale (PSPRS); Total scores range from 0-96 with higher scores indicating more progressed disease

SECONDARY OUTCOMES:
Change in total (10-item) Progressive Supranuclear Palsy Rating Scale (PSPRS) Score | 52 weeks
  Assess the impact of AMX0035 on disease progression as measured by the Progressive Supranuclear Palsy (PSP) Rating Scale (PSPRS); Total scores range from 0-30 with higher scores indicating more progressed disease
Change in MDS-UPDRS Part II Score | 52 weeks
  To evaluate the efficacy of AMX0035 on motor aspects of activities of daily living as measured on the Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-PDRS) Part II; Total scores range from 0-52 with lower scores indicating better function
Frequency of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | 52 weeks
  Safety and tolerability of AMX0035 in participants with PSP

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Amylyx Pharmaceuticals
Locations (62):
- United States (35):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Parkinson's & Movement Disorder Institute, Fountain Valley, California
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Stanford Movement Disorder Center, Palo Alto, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - UC Health Anschutz Outpatient Pavilion Anschutz Medical Campus, Aurora, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - UF Health Dorothy Mangurian Neuroimaging Suite, Gainesville, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Augusta University, Augusta, Georgia
  - Parkinsons and Movement Disorder Center at the Queens Medical Center, Honolulu, Hawaii
  - Northwestern University PD and Movement Disorders Center, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - University of Minnesota, CTSI, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Missouri
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - University of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Veracity Neuroscience, LLC, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Kerwin Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - University of Utah Movement Disorders Center, Salt Lake City, Utah
  - Virginia Commonwealth University Department of Neurology, Richmond, Virginia
- France (7):
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Hopital Caremeau, Nîmes, Gard
  - Groupe Hospitalier Pellegrin - Hôpital Pellegrin, Bordeaux, Gironde
  - CHU de Limoges - Hôpital Dupuytren, Limoges, Haute Vienne
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille Et Vilaine
  - Hopital Roger Salengro - CHU Lille, Lille, Nord
  - Groupe Hospitalier Pitie-Salpetriere, Paris
- Germany (7):
  - Universitaetsklinikum Duesseldorf AoeR, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Krankenhaus Agatharied, Hausham, Bavaria
  - Klinikum der Universität München, Munich, Bavaria
  - Paracelsus-Elena-Klinik Kassel, Kassel, Hesse
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Asklepios Fachklinikum Stadtroda, Stadtroda, Thuringia
- Italy (6):
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Azienda Ospedale-Università di Padova, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
  - Azienda Ospedaliera Universitaria OO. RR. S. Giovanni di Dio e Ruggi D'Aragona, Salerno
- Spain (7):
  - Hospital de Cruces, Barakaldo, Bizkaia
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari i Politecnic La Fe, Valencia, València
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Undecided